CLINICAL TRIAL: NCT03306875
Title: Impact of Brain Connectome and Personality on Cognitive Rehabilitation in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Ralph H.B. Benedict, Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00001899
Record Dates: First submitted 2017-09-27; First posted 2017-10-11 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; cognitive training; telerehabilitation; personality; Conscientiousness; predict
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cognitive Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Training (Experimental): Individuals will take part in a computer-based cognitive training program. The program is aimed at building attention, processing speed, memory, and executive function.
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Cognitive Training — Individuals will take part in a computer-based cognitive training program. The program is aimed at building attention, processing speed, memory, and executive function.

SUMMARY:
This study aims to apply baseline MRI and neuropsychological measures to predict patient responses to behavioral cognitive rehabilitation. Training will take place over 12 weeks, 1 hour per day, 5 days per week.

The investigator hypothesizes the following:

[1a] The investigator expects that individuals with low baseline Conscientiousness will experience a lower magnitude of overall cognitive improvement following rehabilitation

1. b] The investigator expects the impact of Conscientiousness on fidelity of rehabilitation will in part be moderated by individual differences in program adherence and executive function
2. a] The investigator expects that individual differences in structural and functional connectome disturbances will in part explain differences in participant responses to cognitive rehabilitation.

This study will also serve to supplement the sample of participants for the current IRB approved study ((IRB: 603069, Title: A case-control, 5-year follow-up study of cardiovascular, environmental and genetic risk factors for disease progression in patients with multiple sclerosis.

DETAILED DESCRIPTION:
The participant will be asked to make a total of two (2) visits, approximately 90 days apart. Each visit will involve: neuro-performance testing, and self-report questionnaires. Each study visit is expected to take approximately 1-2 hours. Between the two visits, the participant will be asked to complete a 12 week, computer-based cognitive training program. This includes 1 hour of training each day for 5 days each week.

On Visit 1, the participants will undergo a full battery of neuro-performance tasks including tests and questionnaires that will measure their memory, thinking speed, fatigue, and personality. This visit is expected to take approximately 1-2 hours. The participants will be also asked to have a close friend or family member to complete similar surveys. A self-addressed envelope containing these questionnaires will be provided to take home with them. The participant will need to pass it onto a close friend or family member to be completed and mailed back.

In addition, the participant will be asked to take part in the 12 week computerized cognitive training program. This can be done at home, or anywhere the participant has access to a computer and internet. This cognitive training has been shown to improve cognitive performance in people with multiple sclerosis. The training involves a variety of interactive exercises which adapt to their abilities. The participants will need complete 1 hour of training each day, for 5 days each week.

At 90 days, the participant will return for the 1-2 hours' follow-up visit where they will complete the same cognitive testing and questionnaires which they had completed during visit 1.

All study visits will take place at Buffalo General Hospital. All of the procedures described above will be performed by a trained member of the research team as part of the research study.

If an individual is ineligible for participation, their screening information will be discarded (i.e., shredded). If participants are deemed eligible (either in person or over the phone), they will be scheduled to come in to the hospital for neuropsychological testing. Written consent will be obtained prior to administration of tests. As part of the consent process, participants will be asked for permission to use any data collected as part of the screening process as well.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* males and females above age 18
* fluent in English
* education >9 years

Additional inclusion criteria for MS patients are as follows:

* Clinically definite MS diagnosis
* Expanded Disability Status Scale (EDSS) ≤ 6.5
* MS patients must be relapse-free and stable from the time of their MRI acquired for the CEG-MS study
* Willing and able to comply with the study procedures for the duration of the trial

Exclusion Criteria:

* history of serious medical or psychiatric illness (other than MS in the patient group) that may affect cognitive functioning
* color-blindness
* history of developmental disability
* past or current alcohol or substance dependence
* History of major depressive disorder, bipolar disorder, or psychotic disorder predating the onset of MS
* History of traumatic brain injury as defined by trauma causing loss of consciousness or transient post-traumatic or retrograde amnesia exceeding 5 min
* Other pathology related to MRI abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Impact of Conscientiousness on Cognitive Training Outcomes | This outcome will be measured according to changes from baseline cognition to follow-up measures, 12 weeks later (following cognitive rehabilitation)
  The investigator expects baseline Conscientiousness to correlate positively with cognitive gains following rehabilitation.
  Conscientiousness will be measured using the NEO-Five Factor Inventory (NEOFFI). All scores for personality testing will be converted to age-corrected t-scores for final analysis. These are therefore standardized values without units.
Cognitive Training Outcomes | This outcome will be measured according to changes from baseline cognition to follow-up measures, 12 weeks later (following cognitive rehabilitation)
  Cognitive gains will be measured according to differences between baseline and followup testing for the following tests of cognition.
  * Brief Visuospatial Memory Test (BVMT). This is a test of visual and spatial learning and memory.
  * California Verbal Learning Test (CVLT). This is a test of verbal learning and memory.
  * Symbol Digit Modalities Test (SDMT). This is a test of visual information processing speed.
  All scores for cognitive testing will be converted to age-corrected t-scores for final analysis. These are therefore standardized values without units.

SECONDARY OUTCOMES:
Moderating role of executive function | 12 weeks, as above
  The investigator will assess whether baseline scores of executive function moderate the impact of Conscientiousness on cognitive training.
  Executive function will be reported according to scores on the following tests.
  * Delis-Kaplan Executive Function System (D-KEFS) Tower Test.
  * D-KEFS Sorting Test.
  * Elithorn Perceptual Maze Test (EPMT). All scores for executive function will be converted to age-corrected t-scores for final analysis. These are therefore standardized values without units.
Moderating role of program adherence | 12 weeks, as above
  The investigator will assess whether daily program adherence is a moderates the impact of Conscientiousness on cognitive training. Daily program adherence will be measured according to days and hours spent on cognitive training exercises.
Impact of baseline brain connectivity on cognitive rehabilitation outcomes | 12 weeks, as above
  The investigator will assess whether individual differences in structural and functional connectome disturbances in part explain differences in participant responses to cognitive rehabilitation.
  In order to address outcome number 5, white matter tract disruption will be characterized in order to determine how structural networks are impacted by white matter lesions. Tract disruption will be reported as the proportion of tracts normally connecting pairs of gray matter brain regions which are disrupted by lesions. These will therefore be reported as percent values.

CONTACTS AND LOCATIONS:
Locations (1):
- Jacobs Comprehensive Multiple Sclerosis Treatment and Research Center, Buffalo, New York, United States

DOCUMENTS (3):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03306875/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03306875/SAP_001.pdf
  • Informed Consent Form (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03306875/ICF_002.pdf